CLINICAL TRIAL: NCT00891397
Title: Pregabalin vs. Placebo as an Add on for Complex Regional Pain Syndrome of the Upper Limb Managed by Stellate Ganglion Block
Brief Title: Pregabalin Versus Placebo as an Add on for Complex Regional Pain Syndrome (CPRS) of the Upper Limb Managed by Stellate Ganglion Block (The PREGA Study)
Acronym: PREGA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit patients
Sponsor: McMaster University (Other)
Collaborators: Pfizer (Industry); Hamilton Health Sciences Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 07-181
Record Dates: First submitted 2009-04-28; First posted 2009-05-01 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Complex Regional Pain Syndromes
Keywords: CPRS; stellate ganglion block; pregabalin; pain; Type I
MeSH Terms: conditions — Complex Regional Pain Syndromes; Pain | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Pregabalin group is made up of 20 patients. Patients will receive 150mg/day in two divided does. The patients will be assessed weekly and the dose can be increased to 300mg/day, if the patient does not report any decrease in pain. The following week the dose may be increased to 600mg/day if once again the patient reports no decrease in pain. This is also the maximum permissible does that will be given to the patient. If patient reports any side effects then the dose can be decreased once. The time period of 2 to 5 weeks will be the dose adjustment period. After which the drug maintenance period extends from week 5 to 12. All doses will be given in two divided doses/day.
  Interventions: Drug: Pregabalin
- 2 (Placebo Comparator): Ten patients will be be in the placebo group.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Pregabalin — Dose of 150mg/day divided in two doses. Increased to 300mg/day then to 600mg/day, always divided in two doses for the day.
  Other Names: Lyrica
  Arms: 1
Other: Placebo — Sugar pill
  Arms: 2

SUMMARY:
The purpose of this study is to assess the efficacy of pregabalin in patients with complex regional pain syndrome Type I and to determine whether it provides clinically significant pain relief and whether it improves functioning of the upper limb.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with CRPS Type I as per the IASP (International Association for the Study of Pain) criteria which states presence of an initiating noxious event, or cause for immobilization
* Evidence at some point of swelling, color change, hot/cold/sweaty sensation and no other condition which can account for the pain and dysfunction of the upper limb
* Men or women between ages 18-65 year old
* Women should not be pregnant or breast feeding
* No change in treatment for 4 weeks prior to recruitment
* Pain scores of 4/10 on a verbal analogue scale

Exclusion Criteria:

* Patients with a neurologic disorder unrelated to CRPS
* Patients who are already on pregabalin
* Patients with renal impairment whose creatinine clearance is less than 60 ml/min
* Patients with congestive heart failure who are also diabetic and taking thiazolidinedione medication like rivoglitazone
* Unstable psychiatric history
* Patients with another problem with equal or worse pain
* Unstable medical condition

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2007-11; Primary Completion 2010-01 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Pain relief assessed by an observer blinded to group allocation with daily pain scores and assessed weekly. | Three months

SECONDARY OUTCOMES:
Functional disability assessed by an observer blinded to group allocation. Patient rated wrist and hand evaluation form. | Three months

CONTACTS AND LOCATIONS:
Overall Officials: Norman Buckley, MD, Principal Investigator — Hamilton Health Sciences Corporation
Locations (1):
- Hamilton General Hospital, Hamilton, Ontario, Canada

REFERENCES:
- [Background] Freynhagen R, Strojek K, Griesing T, Whalen E, Balkenohl M. Efficacy of pregabalin in neuropathic pain evaluated in a 12-week, randomised, double-blind, multicentre, placebo-controlled trial of flexible- and fixed-dose regimens. Pain. 2005 Jun;115(3):254-263. doi: 10.1016/j.pain.2005.02.032. Epub 2005 Apr 18. PMID 15911152